CLINICAL TRIAL: NCT05429840
Title: A Two-part, Single Dose, Randomized, Single Blinded, Placebo Controlled, Phase I Study to Assess the Safety and Pharmacokinetics of Oral MT1980 in Healthy Volunteers When Dosed in the Fasted State
Brief Title: Safety & PK of Single Doses of MT1980
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Monument Therapeutics Limited (Industry)
Collaborators: ICON plc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PCD101; 2022-000252-11 (EudraCT Number); MUT21622-21622X (Other: Cinical Research Organisation)
Record Dates: First submitted 2022-06-16; First posted 2022-06-23 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Neuroinflammatory Response
Keywords: pharmacokinetics; neuroinflammation
MeSH Terms: conditions — Neuroinflammatory Diseases

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Part 1: Open Label Part 2: Blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Part 1 MT1980 (Experimental)
  Interventions: Drug: MT1980
- Part 1 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2 MT1980 Dose Level 1 (Experimental)
  Interventions: Drug: MT1980
- Part 2 MT1980 Dose Level 2 (Experimental)
  Interventions: Drug: MT1980
- Part 2 Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MT1980 — single dose
  Arms: Part 1 MT1980; Part 2 MT1980 Dose Level 1; Part 2 MT1980 Dose Level 2
Drug: Placebo — single dose
  Arms: Part 1 Placebo; Part 2 Placebo

SUMMARY:
MT1980 is being developed as a treatment for neuroinflammation (an inflammatory response in the brain and/or spinal cord). Much research has focused on the central role of neuroinflammation in the pathogenesis of many conditions relating to the CNS, including eg, traumatic brain injury, stroke, Alzheimer's disease, post-operative cognitive decline (POCD)/perioperative neurocognitive disorder, and now even long-term cognitive side effects from severe acute respiratory syndrome corona virus 2 (SARS-CoV-2). Current anti-inflammatories do not easily cross the blood-brain barrier from the systemic circulation to the brain, making neuroinflammation a difficult condition to treat.

This will be a Phase 1, single dose, randomized, placebo-controlled study in healthy subjects. The study will provide information on the safety of MT1980, the systemic bioavailability of the active drug, and levels of the active drug in the CSF. The study will be conducted in two parts. In Part 1, subjects will be randomized to receive a single oral dose of MT1980 or placebo in a parallel design. An interim PK and safety data analysis will be performed after Part 1 prior to dose selection in Part 2. In Part 2 subjects will be randomized to receive either placebo or a single oral dose of MT1980 at one of 2 strengths in a parallel design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers with good physical and mental health
* Body Mass Index 18 to 30 kg/m2
* Men & women of child-bearing potential must agree to use adequate contraception
* Willing & able to provide written informed consent and to communicate and participate in the study

Exclusion Criteria:

* Clinically significant abnormal biochemistry, haematology, urinalysis results
* Results of screening liver function or kidney function tests outside of normal ranges
* Heavy daily smoking or use of nicotine containing substances

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-04 (Actual); Study Completion 2022-10-04 (Actual)

PRIMARY OUTCOMES:
Treatment-related adverse events | Day 1 to Day 11
  Descriptive statistics comparing MT1980 & placebo following a single dose of study drug. Number of subjects, number of events and severity of events to be reported

SECONDARY OUTCOMES:
Systemic bioavailability of MT1980 | 72 hours post dose
Level of MT1980 in CSF | up to 7 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Principal Investigator, Principal Investigator — Icon Early Development Services
Locations (1):
- Icon Early Development Services, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No